CLINICAL TRIAL: NCT04731597
Title: Drug Interactions and Hip Fracture Risk in Older Adults
Status: Completed | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, CRISTINA MARIA ELIZONDO, Principal Investigator, Hospital Italiano de Buenos Aires
Other Study IDs: 3804
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Drug Interactions

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases with hip fracture: Patients afiliated to a HMO Plan de Salud Hospital Italiano who presented hip fracture between 2014 and 2019
  Interventions: Drug: drug interaction
- controls without hip fracture: Patients afiliated to a HMO Plan de Salud Hospital Italiano without hip fracture between 2014 and 2019
  Interventions: Drug: drug interaction

INTERVENTIONS:
Drug: drug interaction — when two drugs are taken together

SUMMARY:
Older people are in great risk of hip fracture for multiple reasons. Also they often are on medications for medical conditions. Hip fracture risk increases in relation to some medications. When older peoples take 2 or more medications they are in increase risk of hip fracture.

DETAILED DESCRIPTION:
In this study the investigators describe medication intake profile and identify older people risk of hip fracture in relation to their medication when they are taken together.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated patients to the HMO Plan de Salud Hospital Italiano at least 6 months affiliated.

older than 64 years old

* affiliated between 01/07/2014 al 31/12/2019.

Exclusion Criteria:

* Pathological Hip fracture
* bilateral elective hip replacement previous study period

Min Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cases:
  * Affiliated patients to the HMO Plan de Salud Hospital Italiano at least 6 months affiliated.
  * older than 64 years old. affiliated between 01/07/2014 al 31/12/2019.
  * traumatic hip fracture. controls:
  * Affiliated patients to the HMO Plan de Salud Hospital Italiano at least 6 months affiliated. * older than 64 years old.
  * affiliated between 01/07/2014 al 31/12/2019.
  * without traumatic hip fracture.
Sampling Method: Probability Sample
Enrollment: 9721 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
hip fracture | 1 year
  non pathological hip fracture

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Italiano de Buenos Aires, CABA, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No